CLINICAL TRIAL: NCT04108364
Title: Voice Adaptive Training for Adults With Aphasia
Brief Title: Voice Adaptive Tablet-Based Naming Treatment for Adults With Aphasia
Acronym: VoiceAdapt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Toronto (Other); Technische Universität Berlin (Other); AIT Austrian Institute of Technology GmbH (Other); Nurogames GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MYB155164
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-01

CONDITIONS: Aphasia
Keywords: aphasia; anomia; rehabilitation; speech-language pathology; mobile applications; language therapy; stroke; stroke rehabilitation
MeSH Terms: conditions — Aphasia; Anomia; Stroke

STUDY DESIGN:
Intervention Model Description: two arm, randomized, waitlist-controlled, crossover group design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VoiceAdapt Intervention (Experimental): PWA who train with VoiceAdapt app
  Interventions: Behavioral: Voice adaptive training for aphasia
- No Intervention (No Intervention): PWA who are on the waitlist and not training with VoiceAdapt app

INTERVENTIONS:
Behavioral: Voice adaptive training for aphasia — Training with the VoiceAdapt tablet-based therapy app 25 hours (1 hr/day x 5 days/week x 5 weeks)
  Arms: VoiceAdapt Intervention

SUMMARY:
Rising life expectancy is leading to a rising incidence of strokes worldwide. Approximately one third of people who had a stroke live with a communication disorder, aphasia, which is associated with the largest negative relationship to quality of life. In chronic stages, people with aphasia (PwA) often do not receive any rehabilitation, despite treatment being shown to significantly reduce impairment. In contrast to existing computerized aphasia treatment, VoiceAdapt is an innovative and motivating application for PwA that provides adaptive and context-aware training lessons via speech interaction on the mobile device. A user-centred design process and motivational gamification ensure long-term engagement in training. Through providing an autonomously usable and low-cost tool, VoiceAdapt will positively affect PwA's self-esteem and social inclusion, leading to higher quality of life.

DETAILED DESCRIPTION:
Purpose:

The purpose of the study proposed in this ethics application is to examine the impact of an adaptive speech-language treatment app, created using principles of user-centred design, on language and communication outcomes of people with aphasia (PwA) within a randomized controlled trial.

Background:

Nearly one third of individuals who have a stroke will present with aphasia, a communication impairment that affects the ability to speak, understand, read and write. People with aphasia (PwA) have been shown to demonstrate more limitations in their participation in daily activities, lower quality of life and a higher incidence of depression relative to post-stroke individuals without aphasia, even when other factors such as physical ability, social support and well-being were similar.

The overall goals of the VoiceAdapt research project are to: 1) conduct a needs survey with PwA and speech-language pathologists (SLPs); 2) develop an app employing a user-centred design process; and 3) conduct a randomized controlled trial. Using user-centred design, end users and stakeholders (PwA, therapists and formal/informal caregivers) will be engage din a needs survey during the technology development process. Outcomes will be analyzed to elaborate implications for decision makers as to how to implement such adaptive training environments in stroke rehabilitation. This aspect of the research (i.e., Goals 1 & 2) will be carried out by consortium members in Austria and Germany. Only the randomized controlled trial (Goal 3), which is the subject of the present application, will be conducted at the University of Alberta and the University of Toronto.

PwA will be provided with a personalized speech-language treatment app (i.e., on a tablet), which automatically adapts the exercises to the users' actual skill level. Individual learning progress of PwA will be supported by personalized and gamified training elements to achieve higher compliance and adherence to the exercises. As a primary outcome, the adaptive assistive technology will examine language performance related to the specific intervention of the personalized speech-language treatment app. Additional objectives will examine the change in the overall language and communication functioning of PwA; the well-being and quality of life of PwA and their caregiver's perception of communication effectiveness after intervention with the treatment app.

The research will be carried out by the VoiceAdapt Consortium, which brings together the resources of five participating international institutions. Research partners have expertise in the fields of technology/e-health and graphical design skills (Nurogames, NG), personalization and adaptvitiy (Technical University of Berlin, TUB), user-centred design and gamification/persuasion (Austrian Institute of Technology, AIT), and clinical research and intervention studies (University of Toronto, UoT; University of Alberta, UoA).

Research Methods/Procedures:

Researchers at the University of Alberta and University of Toronto will be the primary investigators of the randomized controlled trial (RCT) portion of the VoiceAdapt Project. The RCT will involve 80 PwA in total across University of Alberta and University of Toronto sites.

Design of the RCT: The RCT will be a two arm, randomized, waitlist-controlled, crossover group design. In Phase 1, PWA randomized to the intervention group will train with VoiceAdapt. The control group will be a waitlist treatment-deferred group. In Phase 2, the control group will train with VoiceAdapt. The randomization of participants will be achieved by computer-generated assignment.

Participants: All participants will have suffered a left hemisphere stroke, be at least 6 months post-onset, and will have aphasia as defined by performance on the Western Aphasia Battery - Rev. (Aphasia Quotient greater than or equal to 30, with a prominent verbal expression impairment), but type of aphasia will not be an inclusion criterion. Participants will speak English as their primary language, pass screenings of visual perception, hearing and basic cognitive functioning and be willing to commit to participation for the study duration.

Intervention: Each intervention phase will last for 5 weeks. During this period, participants in the experimental condition will be asked to do speech language tasks 5 days a week for 60 minutes via the VoiceAdapt app (intervention group). The control group will not be engaged in any one on one speech therapy during the first intervention phase (Phase 1). During the second intervention phase (Phase 2), the control group will participate in training with the VoiceAdapt app (60 minutes/day x 5 days/week) and the intervention group from Phase 1 will crossover into receiving no treatment. Research staff will check in with individuals in the intervention group on a weekly basis to monitor and adjust treatment exercises. Research staff will check in with participants in the control group twice during their respective control phase.

Outcome Measures: In line with the recommended core outcome measures for aphasia research (Wallace et al., 2019), participants in both groups will be tested before and after each condition on the following measures: the primary outcome measure will be the Boston Naming Test (BNT) to measure naming; secondary outcome measures will be: Western Aphasia Battery-Revised (WAB-R); Stroke and Aphasia Quality of Life Scale (SAQOL-39) to measure quality of life; and Communication Effectiveness Index (CETI) to measure the person with aphasia and the partners' perception of the participant's communication. In addition to these measures, the Situational Motivation Scale (SIMS) and an end of study questionnaire will be provided to all participants.

Plan for Data Analysis:

The primary analysis will be a one-sided hypothesis test of the null hypothesis of the change in naming on the Boston Naming Test (BNT) from baseline to week 6, tested at the 0.1 level of significance. The observed change on the BNT as well as the baseline, 6 week and follow up values will be summarized for each group as means and standard deviations. Secondary outcomes will be summarized using means (SD), medians (IQR) or proportions (CI), and analyzed using t tests, as appropriate. All analyses will be presented in aggregate.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 6 months post onset of a single stroke in the left hemisphere
2. have aphasia of mild to moderate severity (Aphasia Quotient ≥ 30 on WAB--R) with a prominent verbal expression impairment.
3. pass screenings of visual perception (BORB), hearing (pure tone screening with portable audiometer), and basic cognitive functioning (Raven's Coloured Progressive Matrices)
4. speak English as a primary language.
5. be willing to commit to participation for study duration

Exclusion Criteria:

* Currently participating in individual (one-on-one) speech-language therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Change in naming on the Boston Naming Test (BNT) | baseline; 7 weeks; 13 weeks
  Naming performance (out of 60) on the BNT

SECONDARY OUTCOMES:
Change in Aphasia Quotient on the Western Aphasia Battery-Revised (WAB-R) | baseline; 7 weeks; 13 weeks
  Score on the Aphasia Quotient (out of 100) portion of the WAB-R to measure general communication/language
Change in score on the Stroke and Aphasia Quality of Life Scale (SAQOL-39) | baseline; 7 weeks; 13 weeks
  Mean score (range = 1-5) on the SAQOL-39 to measure overall quality of life; higher scores indicate higher quality of life
Change in score on the Communication Effectiveness Index (CETI) | baseline; 7 weeks; 13 weeks
  Mean score (out of 100) of items on the CETI (16 questions) to measure partners' perception of the participant's communication; higher scores indicate higher communicative effectiveness

OTHER OUTCOMES:
Situation Motivation Scale (SIMS) score | 7 weeks; 13 weeks
  mean score (range = 1-7) on items constituting 4 subscales of SIMS (intrinsic motivation, identified regulation, external regulation, amotivation) will be used to measure participants' motivation while engaging in training; higher scores indicate higher levels of construct measured

CONTACTS AND LOCATIONS:
Overall Officials: Esther S Kim, PhD, Principal Investigator — University of Alberta; Elizabeth Rochon, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim ES, Laird L, Wilson C, Bieg T, Mildner P, Moller S, Schatz R, Schwarz S, Spang R, Voigt-Antons JN, Rochon E. Implementation and Effects of an Information Technology-Based Intervention to Support Speech and Language Therapy Among Stroke Patients With Aphasia: Protocol for a Virtual Randomized Controlled Trial. JMIR Res Protoc. 2021 Jul 2;10(7):e30621. doi: 10.2196/30621. PMID 34255727